CLINICAL TRIAL: NCT06948227
Title: Effect Of Social Robots On Motivation And Participation In Activities Of Daily Life Training In Cerebral Palsy
Brief Title: Effect Of Social Robots In Cerebral Palsy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Collaborators: Yeditepe University (Other)
Responsible Party: Principal Investigator, Hale Nur Baş, Occupational Therapist, Medipol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMU-ERG-HNB-01; 123E355 (Other Grant/Funding Number: The Scientific and Technological Research Council of Turkey)
Record Dates: First submitted 2025-04-21; First posted 2025-04-29 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Cerebral Palsy (CP)
Keywords: cerebral palsy; nao; occupational therapy
MeSH Terms: conditions — Cerebral Palsy | interventions — Activities of Daily Living

STUDY DESIGN:
Intervention Model Description: Two groups as Daily Living Activities (ADL) Training Program and Social Robot Application Group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Social Robot Application Group (Experimental): The negatively affected characteristics of children with Cerebral Palsy will be determined by the occupational therapist together with their families. Activities that they cannot do in daily life will be implemented using the Social Robot Nao within the occupational therapy application to improve their upper extremity skills and motivation.
  Interventions: Other: Social Robot Application
- Daily Living Activities (ADL) Training Program Group (Active Comparator): The negatively affected characteristics of children with cerebral palsy will be determined by the occupational therapist together with their families. Occupational therapy will be applied to the activities they cannot do in daily life by developing their upper extremity skills and motivation.
  Interventions: Other: Daily Living Activities (ADL) Training Program

INTERVENTIONS:
Other: Daily Living Activities (ADL) Training Program — After the 1st assessment, activities that the investigators frequently use in daily life such as eating and brushing our teeth and activities that are appropriate for the age group of the participants and that affect their participation such as throwing a ball or playing games will be implemented with the therapist for 6 weeks. During the session, the therapist will provide practical training so that the participants can do the activities correctly and will provide a demonstration of the activity, observe whether the child compensates while performing the movements during all these activity steps and will make corrections for the movements that he/she compensates for. At the same time, the therapist will give reinforcing verbal affect for the activity skills that the participants do correctly in order to increase their motivation during the session. The 2nd Assessment will be made at the end of the 6th week in order to analyze the change during the 6-week period.
  Arms: Daily Living Activities (ADL) Training Program Group
Other: Social Robot Application — The basic daily life activities that the Social Robot can perform, such as eating and brushing teeth, and the ball throwing activity that affects their participation, will be coded into the robot by engineers. 1. The evaluations will be applied as in the other group, and occupational therapy sessions for upper extremity skills will be applied with the Social Robot Nao accompanied by a therapist for 6 weeks. In this group, the robot will show the selected activities to the children according to the activity application steps during the session and then ask the child to apply them. The verbal feedback that the Social Robot Nao will use will be determined and applied by the therapist. At the end of the 6th week, the second evaluations will be made and the 6-week developments of the participants in this group will be analyzed. Each session will be applied once a week for 40 minutes.
  Arms: Social Robot Application Group

SUMMARY:
The aim of this study is to compare the motivation of the participants, upper extremity skills and daily living activity skills of classical occupational therapy practices in children diagnosed with cerebral palsy with therapy practices using Social Robot Nao in addition to classical occupational therapy practices.

DETAILED DESCRIPTION:
Social Robots are technological developments that are used very frequently, especially in sectors such as education, health and industry, and whose use is increasing day by day, providing services by providing human-robot interaction in various application areas. This study aims to support upper extremity skills in children diagnosed with cerebral palsy through interaction, to increase participation by teaching daily living activities, and to examine the effects of this therapy in the long term. With the social robot, occupational therapists and physiotherapists will be prevented from suffering from burnout syndrome by increasing their efficiency in therapy. One of the aims is to increase motivation in therapy through interaction with the social robot and to maintain the positive effects of therapy in the long term.

Cerebral palsy is defined as a permanent movement and posture disorder that occurs with a non-progressive lesion in the developing fetal and newborn brain and causes activity limitation. Cerebral Palsy is classified as spastic, dyskinetic, ataxic according to movement disorder, and as diplegia, quadriplegia, triplegia and hemiplegia according to the affected body part. In hemiplegic type cerebral palsy, which is the most common type in which one side of the body is used more than the other in classification according to body part, the upper extremity is generally affected more than the lower extremity. In the classification according to movement disorders, the most common one is unilateral spastic cerebral palsy, which negatively affects the ability to perform daily living activities, especially due to difficulties in grasping skills. Shoulder adduction-internal rotation contracture, elbow flexion contracture, wrist flexion-pronation contracture are the most common symptoms, especially in the upper extremity, but factors such as the patient's existing spasticity, affected muscle and age may cause changes in symptoms. Therefore, upper extremity movement analyzes are complex. Children with cerebral palsy often have difficulty with activities that the investigators need in daily life, such as grasping and manipulating objects. This difficulty occurs very often, especially when doing activities that require fine motor skills and the use of both hands (bimanual actions). The aforementioned bimanual actions are important in performing daily living activities such as buttoning shirts, tying shoelaces, opening bottle caps, and using cutlery, which require advanced fine motor skills and a large number of tasks and variety.

In recent years, new technological advances in walking, balance and upper extremity skill rehabilitation have been made available to patients with cerebral palsy. One of these is the social robot Nao, which teaches upper extremity motor functions required for daily living activities in children with cerebral palsy through imitation, and is known to be used successfully in rehabilitation. Social robots, which provide social communication by interacting with users, have been frequently used as assistants in the rehabilitation process in recent years. These social robots benefit from their physical, social and emotional characteristics to both progress in therapies and maintain commitment as well as effective communication. Thanks to these characteristics, therapies are long-lasting. Social robots are specifically designed to sustain and promote the effectiveness of therapies and education in children. The social robot Nao is more affordable than other types of robots and has a variety of functionality, making it the most frequently preferred choice in therapies. There are studies in the literature on the use of the social robot Nao in therapies to improve motor skills in daily life activities in children diagnosed with cerebral palsy. It has also been used previously in upper extremity rehabilitation and has proven to be a tool in teaching activities through imitation.

Although there are many studies in the literature on the use of social robots in rehabilitation, the examination of their effects on motivation and participation in these rehabilitation programs has been insufficient. The aim of this study is to teach upper extremity skills to children diagnosed with cerebral palsy through imitation activities using a social robot and to examine the effects on their motivation and participation. This study is original in that it adds a social robot to occupational therapy sessions and examines the effects of participation and motivation on children with cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

* Children with levels I-III according to the Gross Motor Function Classification System (GMFCS),
* Children with levels 1-3 according to the Manual Ability Classification System (MACS),
* Children with levels 0-2 according to the Modified Ashworth Scale,
* Children with levels 1-2 according to the Communication Function Classification System (CFCS),
* Children between the ages of 4-12,
* Children with cerebral palsy will be included in the study.

Exclusion Criteria:

* Children who have not had any orthopedic surgery affecting the upper extremity in the last year
* Children who have any epileptic findings
* Children who have received botox in the last 6 months will be excluded from the study.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-10-25 (Estimated)

PRIMARY OUTCOMES:
Quality of Upper Extremity Skills Test (QUEST) | six weeks
  This scale will be applied to analyze the changes in the upper extremity skills of the participants. In this scale, the investigators put a check mark on the skill that the participant can do. The investigators cross out the skill that the participant cannot do, and write NT for the skill that cannot be tested. This scale has dissociated movements, grasps, wight bearing and protective extansion.The higher the total score, the more advanced the skill. There is a separate calculation method for each subsection. In the final stage, to calculate the total score of the test, the scores obtained in each subsection are added up and divided by the number of sections tested [ [(Score A-50)x2 + (Score B-50)x2 + (Score C-50)x2 + (Score D-50)x2] /4 ].
Bimanual Fine Motor Function (BIMF) | six weeks
  This scale will be applied to analyze the changes in the participants' fine motor skills. In this scale, fine motor skills are determined as 5 levels.
  Level I= One hand: manipulates without restrictions. The other hand: manipulates without restrictions or limitations in more advanced fine motor skills Level II= (a) One hand: manipulates without restrictions. The other hand: only ability to grasp or hold (b) Both hands: limitations in more advanced fine motor skills Level III= (a) One hand: manipulates without restrictions. The other hand no functional ability (b) One hand: limitations in more advanced fine motor skills. The other hand: only ability to grasp or worse Level IV= (a) Both hands: only ability to grasp (b) One hand: only ability to grasp. The other hand: only ability to hold or worse Level V= Both hands: only ability to hold or worse

SECONDARY OUTCOMES:
Canadian Activity Performance Scale (COPM) | six weeks
  This scale will be applied to analyze the activities that the participants have difficulty with in their daily lives and to analyze their changes over time. In this scale, parents of children are interviewed and asked to choose five activities that their children cannot do in the subcategories of self-care, productivity and free time. They are then asked to give performance and satisfaction scores to these activities from 1 to 10 (1: I cannot do it at all, 10: I do it extremely well; 1: I am not satisfied at all, 10: I am extremely satisfied). After all score information is noted, the total score is divided by the number of selected activities to obtain the average score. After a certain period of time, parents are asked to score the same activities again, and if the average score between the two dates is over 2 points, it is considered clinically significant.
Pediatric Evaluation of Disability Inventory (PEDI) | six weeks
  This scale will be applied to determine whether the participants can do the activities in their daily lives. In this scale, the sub-parameters of self-care, mobility and social function are scored as 0: cannot do, 1: can do. All scores are then added up for each section.
Pediatric Motivation Scale (PMS) | six weeks
  This scale will be applied to determine the motivation of the participants in therapies. This scale has 19 items and 2 open-ended questions. The 19 items consist of six subsections: Effort/Importance, Interest/Enjoyment, Competence, Relatedness, Autonomy, Value/Usefulness . Each item is scored from 1 to 5 (1: definitely not true, 2: not true, 3: partially not true, 4: partially true, 5: true, 6: definitely true). Items 3, 4, 6, 8 and 18 are scored in reverse. High scores represent high motivation.

CONTACTS AND LOCATIONS:
Overall Officials: Devrim Tarakcı, Associate Professor, Study Chair — Medipol University
Locations (1):
- Dilbade Special Education Rehabilitation Center, Istanbul, Eyupsultan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosenbaum P, Paneth N, Leviton A, Goldstein M, Bax M, Damiano D, Dan B, Jacobsson B. A report: the definition and classification of cerebral palsy April 2006. Dev Med Child Neurol Suppl. 2007 Feb;109:8-14. PMID 17370477
- [Background] Gonzalez JC, Pulido JC, Fernandez F, Suarez-Mejias C. Planning, execution and monitoring of physical rehabilitation therapies with a robotic architecture. Stud Health Technol Inform. 2015;210:339-43. PMID 25991162
- [Background] Calderita LV, Manso LJ, Bustos P, Suarez-Mejias C, Fernandez F, Bandera A. THERAPIST: Towards an Autonomous Socially Interactive Robot for Motor and Neurorehabilitation Therapies for Children. JMIR Rehabil Assist Technol. 2014 Oct 7;1(1):e1. doi: 10.2196/rehab.3151. PMID 28582242
- [Background] Amirova A, Rakhymbayeva N, Yadollahi E, Sandygulova A, Johal W. 10 Years of Human-NAO Interaction Research: A Scoping Review. Front Robot AI. 2021 Nov 19;8:744526. doi: 10.3389/frobt.2021.744526. eCollection 2021. PMID 34869613
- [Background] Liao YH, Lin TY, Wu CC, Shih YN. Can occupational therapy manpower be replaced with social robots in a singing group during COVID-19? Work. 2021;68(1):21-26. doi: 10.3233/WOR-205096. PMID 33459684
- [Background] Cortes-Perez I, Gonzalez-Gonzalez N, Peinado-Rubia AB, Nieto-Escamez FA, Obrero-Gaitan E, Garcia-Lopez H. Efficacy of Robot-Assisted Gait Therapy Compared to Conventional Therapy or Treadmill Training in Children with Cerebral Palsy: A Systematic Review with Meta-Analysis. Sensors (Basel). 2022 Dec 16;22(24):9910. doi: 10.3390/s22249910. PMID 36560281
- [Background] Cacioppo M, Loos A, Lempereur M, Brochard S. Bimanual movements in children with cerebral palsy: a systematic review of instrumented assessments. J Neuroeng Rehabil. 2023 Feb 27;20(1):26. doi: 10.1186/s12984-023-01150-7. PMID 36849971
- [Background] Sakzewski L, Ziviani J, Boyd R. Systematic review and meta-analysis of therapeutic management of upper-limb dysfunction in children with congenital hemiplegia. Pediatrics. 2009 Jun;123(6):e1111-22. doi: 10.1542/peds.2008-3335. Epub 2009 May 18. PMID 19451190
- [Background] Rozaire J, Paquin C, Henry L, Agopyan H, Bard-Pondarre R, Naaim A, Duprey S, Chaleat-Valayer E. A systematic review of instrumented assessments for upper limb function in cerebral palsy: current limitations and future directions. J Neuroeng Rehabil. 2024 Apr 16;21(1):56. doi: 10.1186/s12984-024-01353-6. PMID 38622731
- [Background] Makki D, Duodu J, Nixon M. Prevalence and pattern of upper limb involvement in cerebral palsy. J Child Orthop. 2014 May;8(3):215-9. doi: 10.1007/s11832-014-0593-0. Epub 2014 May 14. PMID 24824566
- [Background] Gutterman J, Gordon AM. Neural Correlates of Impaired Grasp Function in Children with Unilateral Spastic Cerebral Palsy. Brain Sci. 2023 Jul 21;13(7):1102. doi: 10.3390/brainsci13071102. PMID 37509032
- [Background] Chiu HC, Ada L. Constraint-induced movement therapy improves upper limb activity and participation in hemiplegic cerebral palsy: a systematic review. J Physiother. 2016 Jul;62(3):130-7. doi: 10.1016/j.jphys.2016.05.013. Epub 2016 Jun 17. PMID 27323932
- [Background] Paul S, Nahar A, Bhagawati M, Kunwar AJ. A Review on Recent Advances of Cerebral Palsy. Oxid Med Cell Longev. 2022 Jul 30;2022:2622310. doi: 10.1155/2022/2622310. eCollection 2022. PMID 35941906
- [Background] Hunt M, Everaert L, Brown M, Muraru L, Hatzidimitriadou E, Desloovere K. Effectiveness of robotic exoskeletons for improving gait in children with cerebral palsy: A systematic review. Gait Posture. 2022 Oct;98:343-354. doi: 10.1016/j.gaitpost.2022.09.082. Epub 2022 Sep 26. PMID 36306544